CLINICAL TRIAL: NCT06962033
Title: PRIDE III Prison Interventions and HIV Prevention Collaboration
Acronym: PRIDE III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000037393; 2R01DA029910-11A1 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hiv; Opioid Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Aim 1: 100 (60 prison OAT providers, 15 per country) for surveys, 40 prison OAT providers, 10 per country, for NGT) Aim 2: 200 (100 probation clients, 100 prison and probation staff (officers and leadership)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1- Implementation (Experimental): Scale-up Opioid Agonist Therapy (OAT) as HIV prevention in prisons and pre-trial detention centers in EECA for individuals with Opioid Use Disorder (OUD) and link them to community treatment after release using development of NIATx learning collaboratives with prison OAT providers (addiction care specialists or primary care doctors). OAT scale-up data will be collected from each country's national OAT database, as well as administration of survey to prison narcologists.
  Interventions: Behavioral: Opioid Agonist Therapy
- Aim 2- Scale-Up (Experimental): Scale-up OAT as HIV prevention in the newly formed probation system in EECA for individuals with OUD and link them to OAT treatment as part of routine care to align public safety and public health using development of NIATx learning collaboratives with probation and prison officers in Kyrgyzstan, Tajikistan, Moldova, and Georgia. OAT scale-up data will be collected from each member country's national OAT database, and administer a survey to probation officers.
  Interventions: Behavioral: Opioid Agonist Therapy

INTERVENTIONS:
Behavioral: Opioid Agonist Therapy — Opioid Agonist Therapy (OAT) as HIV prevention

SUMMARY:
The primary objective of this research project is to identify barriers to scale-up of Opioid Agonist Therapy (OAT) in the justice systems (prisons and probation) in Tajikistan, Kyrgyzstan, Moldova, and Georgia, and establish a NIATx learning collaborative to scale-up OAT, and analyze scale-up utilizing latent class growth analyses in people who inject drugs (PWID).

DETAILED DESCRIPTION:
Aim 1 consists of the development of NIATx learning collaboratives with prison OAT providers (addiction care specialists or primary care doctors). This aim is an implementation science aim involving the collection of OAT scale-up data from each country's national OAT database, as well as administration of survey to prison narcologists every 6 months.

Aim 2 consists of the development of NIATx learning collaboratives with probation and prison officers in Kyrgyzstan, Tajikistan, Moldova, and Georgia. Investigators will collect OAT scale-up data from each member country's national OAT database, and administer a survey to probation officers every 6 months. Investigators will also observe and interview probation clients and staff using ethnographic methods.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

1. Quantitative surveys for prison OAT providers

   * Being 18 years or older
   * Being currently assigned and working as a probation OAT provider for a probation site
2. ECHO procedures

Aim 2:

1. Quantitative surveys for people in probation

   * Being 18 years or older
   * Screen yes to opioid injection on the online screener questionnaire
   * Currently in probation
2. Quantitative surveys for probation and prison officers

   * Being 18 years or older
   * Being currently assigned and working as a probation or prison officer at a probation site
3. Focus Groups (People in probation)

   * Being 18 years or older
   * Screen yes to opioid injection criteria on the online screener
   * Currently in probation
4. Focus Groups (Probation and prison officers)

   * Being 18 years or older
   * Being currently assigned and working as a probation or prison officer at a probation
   * Has more than 3 months of field experience
   * Works at a probation site within 25 kilometers of an OAT site

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants receiving opioid agonist therapy (OAT) | baseline up to 4 years
  Number of patients receiving opioid agonist therapy (OAT) per OAT site.

SECONDARY OUTCOMES:
Adherence to NIATx protocol | baseline up to 4 years
  Adherence to NIATx protocol: using the NIATx fidelity scale, a 19-item assesment to measure adherence to the NIATx model on a 5-point scale from 1 (No evidence) to 5 (Extensive evidence).

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University
Locations (5):
- Yale University, New Haven, Connecticut, United States
- Alternative Georgia, Tbilisi, Georgia
- AIDS Foundation East-West (AFEW), Bishkek, Kyrgyzstan
- NGO AFI, Chisinau, Moldova
- Institute for International Health and Education (IIHE), Dushanbe, Tajikistan

IPD SHARING:
Plan to Share IPD: No